CLINICAL TRIAL: NCT02004028
Title: An Open Label Window of Opportunity Phase II Study of the FAK Inhibitor Defactinib VS-6063 in Participants With Surgical Resectable Malignant Pleural Mesothelioma.
Brief Title: Window of Opportunity Study of VS-6063 (Defactinib) in Surgical Resectable Malignant Pleural Mesothelioma Participants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decided to discontinue trial to focus on development program next steps
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6063-203
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Mesothelioma; adenoma; Neoplasms, Mesothelial; Focal Adhesion Kinase Inhibitor
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma; Adenoma; Neoplasms, Mesothelial | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VS-6063 (defactinib) (Experimental): Administered orally (BID) for 12, 21 or 35 days (+/- 2 days)
  Interventions: Drug: VS-6063

INTERVENTIONS:
Drug: VS-6063
  Other Names: defactinib

SUMMARY:
This is an open label neoadjuvant (treatment with VS-6063 prior to mesothelioma surgery) study in subjects with malignant pleural mesothelioma who are eligible for surgery. Subjects will receive VS-6063 (defactinib) 400 mg twice daily for 12, 21, or 35 days or 100 mg formulation twice daily for 21 days. Pre- and post-treatment biopsies and blood samples will be collected. The purpose of this study is to assess biomarker responses from tumor tissue. The safety, pharmacokinetics, and tumor response rate to VS-6063 (defactinib) will be also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant pleural mesothelioma that is not metastatic or unresectable
* Eligible to undergo excisional surgery such as pleurectomy/decortication (P/DC) or any other mesothelioma surgery.
* Localized disease. The malignancy is confined to one affected hemithorax. Mediastinal N2 lymph nodes via cervical mediastinoscopy or EBUS (endobronchial ultrasound) must be negative in order to be eligible
* Grossly normal pulmonary, cardiac function, renal, hepatic hematologic and performance functions
* Male or non-pregnant female
* Age ≥ 18 years of age
* Tissue is required prior to enrollment. If patient was diagnosed outside and tumor tissue is not available, a pleural biopsy for frozen tissue collection is required.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy any time prior to entering the study or at any prior time for mesothelioma. Patients receiving chemotherapy type drugs for benign conditions can participate in this trial
* History of upper gastrointestinal bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug
* Known history of Gilbert's Syndrome or any current hyperbilirubinemia of any cause
* Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug
* Subjects with known infection with human immunodeficiency virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS)
* Subjects with confirmed Hepatitis A, B or C
* Subjects being actively treated for a secondary malignancy or any malignancy within the last 3 years, with the exception of non-melanomatous skin cancer or localized, definitively treated cervical cancer. Men under observation for local prostate cancer are also eligible if they have had stable disease for at least 1 year.
* Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis
* Known history of malignant hypertension
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations which in the opinion of the study investigators would be associated with undue risk of participation in the study
* Use of an investigational drug within 28 days or 5 half-lives prior to first dose.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, M.D., Study Chair — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 VS-6063 (Defactinib): Defactinib 400 mg BID for 12 Days
- Cohort 2: Defactinib 400 mg BID for 35 Days
- Cohort 3: Defactinib 400 mg BID for 21 Days
- Cohort 4: Defactinib 100 mg BID for 21 Days
Period: Overall Study
Arm/Group | Cohort 1 VS-6063 (Defactinib) | Cohort 2 | Cohort 3 | Cohort 4
Started | 10 | 10 | 10 | 5
Completed | 10 | 10 | 10 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Defactinib 400 mg BID for 12 Days
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 5 | 35
Age, Continuous [Median (Standard Deviation); unit: years] | 75.9 (7.69) | 70.6 (9.83) | 71.7 (7.29) | 66.6 (7.50) | 71.9 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 8 | 8 | 8 | 3 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 10 | 9 | 8 | 5 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of pFAK Inhibition in Tumor Tissue
Description: percentage VS-6063 (defactinib)
Time Frame: Cohort 1, From Baseline to Day 12; Cohort 2, From Baseline to Day 35; Cohorts 3, From Baseline to Day 21; Cohorts 3, From Baseline to day 21 day.
Measure: Median (Full Range); unit: percentage of pFAK inhibition in a tumor
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 5
percentage of pFAK inhibition in a tumor | NA [NA to NA] — True baseline sample were not available so post-treatment samples were compared with post-study surgical specimens which was not an accurate baseline measure. | NA [NA to NA] — True baseline sample were not available so post-treatment samples were compared with post-study surgical specimens which was not an accurate baseline measure. | 85.6 [-12.57 to 100] | NA [NA to NA] — Inhibition of tumor FAK was not included in Cohort 4, as per the protocol.

2. Primary Outcome: Evaluate the Pharmacokinetics of VS-6063 (Defactinib), CMax
Description: Maximum observed plasma concentration
Time Frame: 0-24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1: Cohort 1: Defactinib 400 mg BID for 12 days
- Cohort 2: Cohort 2: Defactinib 400 mg BID for 35 days
- Cohort 3 (Fed): Defactinib 400 mg for 21 days
- Cohort 4 (Fasted): Defactinib 100 mg BID for 21 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 (Fed) | Cohort 4 (Fasted)
Number analyzed (Participants) | 10 | 9 | 9 | 5
ng/mL | 1052 (126) | 1052 (126) | 513 (180) | 517 (76)

3. Primary Outcome: Evaluate the Pharmacokinetics of VS-6063 (Defactinib), AUC (Area Under the Curve)
Description: Area under plasma Concentration (AUC) 0 to t
Time Frame: 0-8 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Cohort 2 (Fasted): Defactinib 400 mg BID for 35 days
Arm/Group | Cohort 1 | Cohort 2 (Fasted) | Cohort 3 (Fed) | Cohort 4 (Fasted)
Number analyzed (Participants) | 10 | 9 | 9 | 5
ng*h/mL | 5280 (136) | 5280 (136) | 2753 (198) | 1891 (69)

4. Primary Outcome: Evaluate the Pharmacokinetics of VS-6063 (Defactinib), Median Tmax (h)
Description: Time to Maximum concentration (Tmax)
Time Frame: 0-24 hours
Measure: Median (Full Range); unit: hour
Groups:
- Cohort 1: Cohort 1: Defactinib 400 mg BID for 12 days Cohort 2: Defactinib 400 mg BID for 35 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 (Fed) | Cohort 4 (Fasted)
Number analyzed (Participants) | 10 | 9 | 9 | 5
hour | 1 [1 to 4] | 1 [1 to 4] | 4 [2 to 8] | 1 [1 to 2]

5. Secondary Outcome: Number of Patients With at Least One Adverse Event
Description: Adverse events will be graded by the CTCAE (Common Terminology Criteria for Adverse Events) 4.0 and summarized according to the worst grade observed since the first treatment dose.
Time Frame: Cohort 1, 40 days; Cohort 2, 42 days; Cohort 3, 28 days; Cohort 4, 28 days.
Population: Patients with at least one treatment-related treatment-emergent adverse events
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 400 mg BID for 12 Days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 5
Participants | 10 | 10 | 10 | 5

6. Secondary Outcome: To Evaluate the Tumor Response to VS-6063 (Defactinib)
Description: Modified RECIST criteria for assessment of response in malignant pleural mesothelioma Ann Oncol 2004. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the in the volume of target lesions; Progressive Disease (PD) at least a 20% increase in the volume of target lesions Stable Disease (SD):
  Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter.
Time Frame: Cohort 1, 40 days; Cohort 2, 42 days; Cohort 3, 28 days; Cohort 4, 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 10 | 10 | 5
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 2 | 1 | 0
  Stable Disease | 9 | 4 | 7 | 2
  Progressive Disease | 0 | 3 | 2 | 3
  Non-Evaluable | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Cohort 1, 40 days Cohort 2, 42 days Cohort 3, 28 days Cohort 4, 28 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/10 | 1/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10 | 2/10 | 2/5
Other Adverse Events (participants affected / at risk) | 7/10 | 8/10 | 6/10 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10) | Cohort 3 (N=10) | Cohort 4 (N=5)
International Normalised Ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10) | Cohort 3 (N=10) | Cohort 4 (N=5)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (5) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (4) | 3 (6) | 3 (3) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 2 (2) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning, procedureal complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (5) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT02004028/Prot_SAP_000.pdf